CLINICAL TRIAL: NCT03764644
Title: Web-based Attention Bias Modification Treatment for Childhood Anxiety Disorders: a Randomized, Double-blind, Controlled Trial
Brief Title: Web-based Attention Bias Modification Treatment for Childhood Anxiety Disorders
Acronym: ATTENTIO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim results showed high futility to continue
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Jeroen Legerstee, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S13-11
Record Dates: First submitted 2018-11-30; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Anxiety Disorder; Anxiety Disorder of Childhood; Separation Anxiety Disorder of Childhood, Early Onset; Specific Phobia; Social Anxiety Disorder; Generalized Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders; Phobia, Specific; Phobia, Social; Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: Double blind, sham-controlled, randomized trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined ABMT and CBT (Experimental): 9 sessions of Attention Bias Modification Treatment (dot-probe based of 160 trials) followed by individual Cognitive Behavioral Therapy via FRIENDS program
  Interventions: Behavioral: Combined ABMT and CBT
- Combined Sham ABMT and CBT (Sham Comparator): 9 sessions of Sham Attention Bias Modification Treatment (dot-probe based of 160 trials) followed by individual Cognitive Behavioral Therapy via FRIENDS program
  Interventions: Behavioral: Combined Sham ABMT and CBT

INTERVENTIONS:
Behavioral: Combined ABMT and CBT — ABMT: A trial begins with a fixation cross (+) for 500 ms, immediately followed by a stimuli pair consisting of a neutral and threatening stimulus that is centred horizontally. Stimuli pairs consist of two faces, pictures or words. After presentation of the stimuli pair, a probe (: or ..) always appears on the location of the neutral stimulus. The probe remains on the screen until the participant presses the corresponding key (: or ..), after which the next trial begins. Each session, participants see 160 trials of which 128 trials include one neutral and one threatening stimulus. The remaining 32 trials include a neutral-neutral stimuli pair. CBT: FRIENDS program individual
  Arms: Combined ABMT and CBT
Behavioral: Combined Sham ABMT and CBT — ABMT: A trial begins with a fixation cross (+) for 500 ms, immediately followed by a stimuli pair consisting of a neutral and threatening stimulus that is centred horizontally. Stimuli pairs consist of two faces, pictures or words. After presentation of the stimuli pair, a probe (: or ..) always appears on the location of the neutral stimulus. The probe remains on the screen until the participant presses the corresponding key (: or ..), after which the next trial begins. Of the 160 trials, the probe appears with equal frequency on the location of the neutral and threatening stimulus (128 trials). The remaining 32 trials include a neutral-neutral stimuli pair. CBT: FRIENDS program individual
  Arms: Combined Sham ABMT and CBT

SUMMARY:
Anxiety disorders are the most common childhood psychiatric disorders, with prevalence rates as high as 15% to 20%. Success rates of the first choice treatment strategy (i.e. Cognitive Behavioural Therapy; CBT) are around 50%. Non-response increases the risk for other psychiatric disorders, school dropout, social isolation, alcoholism, and suicide attempts. These negative consequences endorse the urgent need to develop more effective and accessible treatments that enhance effectiveness of current treatment options. A promising new treatment for childhood anxiety disorders is Attention Bias Modification Treatment (ABMT). ABMT is based on evidence that anxiety-disordered individuals selectively allocate their attention toward threatening information (i.e. attention bias). This bias in early and automatic attention processes starts a cascade of subsequent biases in information processing and memory, resulting in heightened anxiety. Attention bias is an underlying mechanism of anxiety. Thus ABMT, which implicitly trains individuals to attend away from threatening information should alleviate anxiety. In contrast to ABMT, CBT explicitly targets later stages of information processing that are under volitional control. Meta-analyses of studies in adults have shown that ABMT indeed results in increased recovery rates and clinically significant changes in anxiety, compared to so-called "sham" attention training (control condition). Imaging studies have shown that ABMT modifies lateral prefrontal cortex activity to emotional stimuli. Despite its promising results, fewer studies have examined ABMT in anxiety-disordered children. The aim of this trial is to enhance treatment effectiveness by combining web-based ABMT with CBT in a large sample of anxiety-disordered children. The primary aim is to compare ABMT-augmented CBT with CBT as monotherapy on recovery rates for anxiety disorders and changes in anxiety. The secondary aim is to compare ABMT with sham attention training on anxiety disorder recovery rates and changes in anxiety. We hypothesize that (1) ABMT-augmented CBT will result in a significantly better treatment success than CBT alone, and (2) ABMT will result in a significantly better treatment success than sham attention training. The design will be a randomized, double-blind, sham-controlled clinical trial.

DETAILED DESCRIPTION:
Anxiety disorders are the most prevalent psychiatric disorders, occurring in among 15% to 20% of children. Cognitive behavioral therapy (CBT) is currently the first-choice treatment for anxiety-disordered children. Despite proven efficacy, almost half of them do not respond, causing prolonged suffering. Children with persistent anxiety have an increased risk for other psychiatric disorders, school dropout, social isolation, alcoholism, and suicide attempts. Another concern is that only a small proportion of anxiety-disordered children actually receive treatment. These negative consequences in combination with the limited accessibility of treatment endorse the urgent need to develop more effective and accessible treatments that can enhance effectiveness of current treatment options.

A newly emerging and promising childhood anxiety treatment is Attention Bias Modification Treatment (ABMT). ABMT is build upon evidence that anxious children tend to selectively focus their attention on threatening information in the context of other non-threatening information, and that attention bias is related to development and maintenance of anxiety disorders. Children with an attention bias scan their environment for potential threat or danger thereby starting a cascade of subsequent processing biases in interpretation and memory, resulting in heightened anxiety.

Hence, as attention bias is an underlying mechanism of anxiety, treatment that diminishes attention bias toward threat in anxiety-disordered individuals should alleviate anxiety. Subsequently, several researchers began to examine the effect of ABMT, which implicitly trains anxiety-disordered individuals to attend away from threat toward neutral information. This is a different approach than CBT, which does not target early and automatic information processes, but addresses later stages of information processing that are under volitional control. Several studies highlighted the potential of ABMT in reducing anxiety levels in adults. A meta-analysis revealed that ABMT in adults produces significantly greater reductions in anxiety than sham control training, with a large effect size in clinical populations. A previous study found that 72% of the adults were free from their primary anxiety disorder after ABMT as compared to 11% after sham attention training, which is far more than CBT. These training effects were maintained at 4-month follow-up. Importantly, ABMT also modifies neural systems that are involved in the control of attention to emotional stimuli, in particular the lateral prefrontal cortex.

Despite the promising results in adults, ABMT has been scarcely examined in children. A few studies demonstrated a significant anxiolytic effect of ABMT, but not of the sham control condition. A major limitation of previous studies is that sample sizes were quite low and that a limited number of training sessions were provided. It has been shown that more training sessions enhance the magnitude of treatment effect. This is the first study that examines the effectiveness of a 9-session web-based ABMT in a large sample of anxiety-disordered children as well as examines the additive effect of web-based ABMT on CBT.

As reviewed above, childhood anxiety disorders are highly prevalent and debilitating, and there is an urgent need for improvement of current treatment strategies. An innovative, but scarcely examined, treatment option for childhood anxiety disorders is ABMT. A randomized, sham-controlled, double-blind trial of web-based Attention Bias Modification Treatment for childhood anxiety disorders will be conducted. One hundred twenty-eight children will be randomly allocated to a 9 session internet-delivered ABMT or sham attention training. The primary aim is to compare ABMT-augmented CBT with CBT as monotherapy on recovery rates for anxiety disorders and changes in anxiety. The secondary aim is to compare ABMT with sham attention training on anxiety disorder recovery rates and changes in anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for participation are children (aged 8 to 16 years)
* Primary diagnosis of separation anxiety disorder,
* Primary diagnosis of generalized anxiety disorder
* Primary diagnosis of specific phobia
* Primary diagnosis of social phobia

Exclusion Criteria:

* IQ below 85
* poor command of the Dutch language
* serious physical disease
* psychosis
* substance abuse
* pervasive developmental disorder
* obsessive-compulsive disorder
* posttraumatic stress disorder
* acute stress disorder
* panic disorder
* major depression
* anxiety medication during treatment
* any concurrent psychotherapy

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Anxiety disorder status | After 3 weeks of ABMT or sham-ABMT
  Free of any anxiety disorder according to the Anxiety Disorders Interview Schedule for Children (ADIS-C)
Anxiety disorder status | After 10 weeks of CBT
  Free of any anxiety disorder according to the Anxiety Disorders Interview Schedule for Children (ADIS-C)
Anxiety disorder status | 6 months follow-up (from last CBT session)
  Free of any anxiety disorder according to the Anxiety Disorders Interview Schedule for Children (ADIS-C)

SECONDARY OUTCOMES:
Number of anxiety disorders | After 3 weeks of ABMT or sham-ABMT, after 10 weeks of CBT, 6 months follow-up
  Number of anxiety disorders according to the Anxiety Disorders Interview Schedule for Children (ADIS-C)
Anxiety symptoms | After 3 weeks of ABMT or sham-ABMT, after 10 weeks of CBT, 6 months follow-up
  Total scale anxiety symptoms according to the Screen for Child Anxiety Related Emotional Disorders (SCARED-R), 69 items, range 0-138, higher score represents more symptoms
Depression symptoms | After 3 weeks of ABMT or sham-ABMT, after 10 weeks of CBT, 6 months follow-up
  Total scale depression symptoms according to the Child Depression Inventory (CDI), 27 items, range 0-54, higher score represents more symptoms
Number of anxiety disorders | After 10 weeks of CBT
  Number of anxiety disorders according to the Anxiety Disorders Interview Schedule for Children (ADIS-C)
Anxiety symptoms | After 10 weeks of CBT
  Total scale anxiety symptoms according to the Screen for Child Anxiety Related Emotional Disorders (SCARED-R), 69 items, range 0-138, higher score represents more symptoms
Depression symptoms | After 10 weeks of CBT
  Total scale depression symptoms according to the Child Depression Inventory (CDI), 27 items, range 0-54, higher score represents more symptoms
Number of anxiety disorders | 6 months follow-up (from last CBT session)
  Number of anxiety disorders according to the Anxiety Disorders Interview Schedule for Children (ADIS-C)
Anxiety symptoms | 6 months follow-up (from last CBT session)
  Total scale anxiety symptoms according to the Screen for Child Anxiety Related Emotional Disorders (SCARED-R), 69 items, range 0-138, higher score represents more symptoms
Depression symptoms | 6 months follow-up (from last CBT session)
  Total scale depression symptoms according to the Child Depression Inventory (CDI), 27 items, range 0-54, higher score represents more symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Legerstee, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC - Sophia Children's Hospital, Rotterdam, South Holland, Netherlands